CLINICAL TRIAL: NCT03837301
Title: Non-exposure Simple Suturing Endoscopic Full-Thickness Resection (NESS-EFTR) With Laparoscopic Sentinel Lymph Node Navigation for EGC (Senorita3-phase 2)
Brief Title: Non-exposure Simple Suturing EFTR (NESS-EFTR) With Laparoscopic Sentinel Lymph Node Navigation for EGC (Senorita3-phase 2)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Chan Gyoo Kim, M.D., National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2018-0162
Record Dates: First submitted 2019-02-03; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NESS-EFTR (Experimental): Non-exposure Simple Suturing Endoscopic Full-Thickness Resection (NESS-EFTR) With Laparoscopic Sentinel Lymph Node Navigation (basin dissection)
  Interventions: Procedure: NESS-EFTR with sentinel lymph node navigation

INTERVENTIONS:
Procedure: NESS-EFTR with sentinel lymph node navigation — Non-exposure Simple Suturing Endoscopic Full-Thickness Resection with sentinel lymph node navigation (basin dissection) for early gastric cancer patients

SUMMARY:
Laparoscopic sentinel lymph node dissection and stomach preserving surgery in early gastric cancer is less invasive method which can increase quality of life. Current stomach preserving surgery after sentinel lymph node dissection produce transmural communication and expose the tumor to the peritoneum during operation. An endoscopic full-thickness resection method with a simple suturing technique that does not expose the gastric mucosa to the peritoneum (non-exposure simple suturing endoscopic full-thickness resection, NESS-EFTR) was recently developed.

This is the phase2 study to identify the efficacy of NESS-EFTR with sentinel node navigation in early gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* single lesion of adenocarcinoma in preoperative endoscopic biopsy
* clinical stage T1N0 in the preoperative evaluation of endoscopy and computed tomography
* tumor size: less than 3cm
* location: 3cm far from the pylorus or cardia
* aged 20 to 80
* ECOG 0 or 1
* patient who signed the agreement
* patient who is suspected to underwent laparoscopy assisted gastrectomy

Exclusion Criteria:

* absolute indication of endoscopic submucosal resection
* inoperable due to poor cardiac, pulmonary function
* pregnant
* having allergic reaction, previous upper abdominal surgery except laparoscopic cholecystectomy, previous radiation therapy to upper abdomen
* diagnosed as malignancy within 5 years except carcinoma in situ of cervix cancer and thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
complete resection rate (%) of tumor | 2 weeks
  the definition of complete resection is 'Tumor exist in single resected piece (en bloc resection) with clear resection margin'.

CONTACTS AND LOCATIONS:
Overall Officials: Chan G Kim, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang, South Korea

IPD SHARING:
Plan to Share IPD: No